CLINICAL TRIAL: NCT01623063
Title: Histomorphometry Analysis in Fertile and Infertile Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Dani Ejzenberg, MD, MD, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EIFMUSP
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Infertility
Keywords: endometrium; infertility; uterus; histeroscopy
MeSH Terms: conditions — Infertility | interventions — Hysteroscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infertile (Experimental): patients from our human reproduction center
  Interventions: Procedure: Hysteroscopy
- Fertile (Active Comparator): patients with comproved fertility
  Interventions: Procedure: Hysteroscopy

INTERVENTIONS:
Procedure: Hysteroscopy — hysteroscopy with guided biopsies
  Other Names: Bettocchi system- Karl Storz; pipelle- cornier

SUMMARY:
To detect similarities and differences in the endometrium of fertile and infertile patients

DETAILED DESCRIPTION:
morphometric and pathologyc analysis of the endometrium in fertile and infertile patients

ELIGIBILITY:
Inclusion Criteria:

* 18 to 41 years old
* regular menses
* infertility over 12 months

Exclusion Criteria:

* previous uterine surgery
* use of contraceptive pills or injections less than 3 months from the inclusion in the study

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
glandular volume | 1 month
  verify the glandular volume in fertile and infertil patients during the implantation window

SECONDARY OUTCOMES:
epitelial surface | 1 month
  to detect differences in the endometrium of fertile and infertile patients

CONTACTS AND LOCATIONS:
Overall Officials: Dani Ejzenberg, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinicas, São Paulo, São Paulo, Brazil